CLINICAL TRIAL: NCT01015898
Title: Short Term Effects of Photodynamic Therapy in Basal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Zohreh Tehranchi-nia, assistant professor of dermatology Shaheed Beheshti Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pdt1; NCT00985830 (Other Grant/Funding Number: skin research center of ShaheedBMU)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma; photodynamic therapy; photo chemotherapy; basal cell epithelioma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BCC, ALA-PDT (Experimental): Patients with histologically proven basal cell carcinoma who were candidates for treatment with ALA-PDT
  Interventions: Radiation: photodynamic therapy

INTERVENTIONS:
Radiation: photodynamic therapy — treatment of bcc with 5_ALA cream 20% topical administration once monthly+ photodynamic therapy (red light) 120 j/cm2 once monthly
  Other Names: PDT 1200L Waldman Medizintechnik, Villengen; Schwenningen, Germany

SUMMARY:
The purpose of this study is to evaluate the efficacy of photodynamic therapy in treatment of Basal cell carcinoma (BCC) and factors that affect response rate.

DETAILED DESCRIPTION:
Background and Aim: Basal cell carcinoma (BCC) is the most common skin cancer .Photodynamic therapy _as a novel , non-invasive therapeutic approach _may be considered a valuable strategy. This study was designed with the aim of the evaluation of efficacy of PDT in treatment of BCC and factors that may affect response rate.

Materials and Methods: This was a clinical trial which was done on 28 BCCs. Patients were treated with ALA-PDT monthly for 1-6 sessions and evaluated for clinical response,cosmetic results and probable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven BCCs

Exclusion Criteria:

* Rodent ulcer
* Morphea type
* ANA +
* History of photosensitivity or photodermatosis or ingestion of phototoxic
* Drugs during last month
* Pregnancy
* Breast feeding
* Age< 18
* History of another therapeutic intervention for bcc during last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zohreh Tehranchi-nia, assist.prof., Principal Investigator — Skin Research Center